CLINICAL TRIAL: NCT00176371
Title: Improvement of Physical Activity and Correction of Body Mass Index in School Children
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Head of the study has left the institution. Study never started.
Sponsor: University of Leipzig (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: school project
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2018-06-29 (Actual); Status verified 2006-09

CONDITIONS: Overweight
Keywords: Physical fitness
MeSH Terms: conditions — Overweight | interventions — Exercise

INTERVENTIONS:
Behavioral: physical exercise

SUMMARY:
There is an increasing incidence of overweight children in Germany, due to a lack of physical activity.

The aim of this study is to improve physical fitness and activity in school children. Two classes in different schools are provided with additional sport lessons over a period of one year.

DETAILED DESCRIPTION:
The increasing incidence of overweight children in Germany is due to a lack of physical activity and intake of unhealthy food. The importance of physical activity for the prevention of cardiovascular diseases in adults was shown in several trials. Therefore we provide additional sport lessons over the period of one year in two defined schools in Leipzig with the aim to improve physical fitness in school children. Two other classes with the -in germany- usual quantity of sport classes served as control classes.

In all classes at the beginning and at the end of the school year blood samples were taken, and a clinical investigation, a coordination test for children and a spiroergometer were performed. Additionally each child had to fill out a questionnaire.

Endurance training is emphasized in the sport lessons.

ELIGIBILITY:
Inclusion Criteria:

* School class

Exclusion Criteria:

* Condition precluding exercise

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2005-07; Study Completion 2006-12

PRIMARY OUTCOMES:
Improvement of maximal oxygen uptake

SECONDARY OUTCOMES:
Change in body mass index

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Schuler, Professor, Principal Investigator — University of Leipzig
Locations (1):
- University of Leipzig, Leipzig, Saxony, Germany

REFERENCES:
- [Derived] Walther C, Mende M, Gaede L, Muller U, Machalica K, Schuler G. [Effects of daily physical exercise at school on cardiovascular risk--results of a 2-year cluster-randomized study]. Dtsch Med Wochenschr. 2011 Nov;136(46):2348-54. doi: 10.1055/s-0031-1292049. Epub 2011 Nov 8. German. PMID 22068444
- [Derived] Walther C, Gaede L, Adams V, Gelbrich G, Leichtle A, Erbs S, Sonnabend M, Fikenzer K, Korner A, Kiess W, Bruegel M, Thiery J, Schuler G. Effect of increased exercise in school children on physical fitness and endothelial progenitor cells: a prospective randomized trial. Circulation. 2009 Dec 1;120(22):2251-9. doi: 10.1161/CIRCULATIONAHA.109.865808. Epub 2009 Nov 17. PMID 19920000